CLINICAL TRIAL: NCT05032573
Title: Reducing Facial Pain With an Olive Oil Enriched Diet: A Feasibility Study
Brief Title: Feasibility of Olive Oil for Reducing Facial Pain of Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB202100950
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive Oil (Experimental): Incorporating 60 mL of olive oil into usual diet and Dietary Guidelines recommendations
  Interventions: Dietary Supplement: Olive oil and Dietary Guideline recommendations
- Control (Active Comparator): Dietary Guidelines recommendations
  Interventions: Other: Dietary Guideline recommendations

INTERVENTIONS:
Dietary Supplement: Olive oil and Dietary Guideline recommendations — 60 mL of olive oil and healthy diet recommendations
  Arms: Olive Oil
Other: Dietary Guideline recommendations — healthy diet recommendations
  Arms: Control

SUMMARY:
This is a 16-week non-blinded, parallel, controlled trial to determine the feasibility and potential efficacy of an olive oil dietary intervention to alleviate facial pain caused by trigeminal neuralgia type 1 (TGN).

DETAILED DESCRIPTION:
Trigeminal neuralgia (TGN) pain is debilitating and unpredictable. Alleviation of intensity or frequency to any degree will improve the quality of life of the individuals affected. Current medical treatments for TGN are often not effective. In some cases, the pain is a result of myelin degeneration. If diet can provide the basic building blocks for myelin regrowth, then the investigators may be able to reduce facial pain by supporting the myelin nerve sheath.

Animal studies have shown that a dietary intervention with olive oil favorably impacts myelin but no human study has been conducted to date. The investigators propose undertaking a feasibility study to determine if a comparable intervention may work in a similar way in humans. If olive oil impacts myelin repair, then pain will be decreased by this dietary intervention and quality of life will be improved. However, it is not known if individuals with TNG will be able to consume a diet relatively high in olive oil. Feasibility will include testing the logistics of distributing the olive oil intervention to the study subjects, incorporation of olive oil into the participants' daily diets, and online/distance monitoring of compliance and reporting of pain intensity, pain frequency, and quality of life. This feasibility study will lay the groundwork for potential future studies examining the efficacy of olive oil on alleviating facial pain caused by TNG and may provide data for a power analysis for a future interventional trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Trigeminal Neuralgia
2. Able to provide written informed consent in English
3. Self-identifying females 18-99 years of age
4. Willing to consume 60 mL (4 tablespoons) of olive oil and accommodating dietary changes, and thereby achieve weight maintenance.
5. Willing to provide information about dietary intake at baseline, at the study midpoint, and at the end of the study to assess dietary changes.
6. Willing to complete online questionnaires associated with the study.
7. Willing and able to provide a valid social security for study payment purposes.
8. Have access to the internet to complete online questionnaires
9. Willing to maintain confidentiality of the Penn Facial Pain Scale

Exclusion Criteria:

1. Do not meet the above criteria.
2. Currently participating in another interventional clinical trial.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Compliance to olive oil intervention | 12 weeks
  Daily olive oil intake in tablespoons per day.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno ML, Percival SS, Kelly DL, Dahl WJ. Daily olive oil intake is feasible to reduce trigeminal neuralgia facial pain: A pilot study. Nutr Res. 2024 Mar;123:101-110. doi: 10.1016/j.nutres.2024.01.005. Epub 2024 Jan 10. PMID 38306883